CLINICAL TRIAL: NCT04211805
Title: Real World Study of Tenofovir Alafenamide Versus Tenofovir Disoproxil Fumarate to Prevent Vertical Transmission of Hepatitis B in Mothers With High Viral Load
Brief Title: Maternal Therapy With TAF Versus TDF to Prevent Vertical Transmission of Hepatitis B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New Discovery LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CN-P919-2020
Record Dates: First submitted 2019-12-06; First posted 2019-12-26 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Hepatitis B, Chronic; Pregnancy Related
Keywords: Chronic Hepatitis B; Pregnancy; Mother to Child Transmission; Vertical Transmission
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide; hepatitis B hyperimmune globulin; Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Arm (A) TAF Group Comprised of Patients from 11 Centers.: 225 consecutive patients will be treated with local standard of care. The antiviral drug Tenofovir Alafenamide (TAF) will be used to treat highly viremic chronic hepatitis B mothers from the gestational week 24-28 of pregnancy to delivery of infant at eleven centers across the People's Republic of China (PRC). Infants will receive hepatitis B vaccine plus HBIg at birth (within 12 hours) and additional hepatitis B vaccine at the age of week 4 and week 24.
  Interventions: Drug: Tenofovir Alafenamide 25 MG for arm (A)
- Arm (B) TDF Group Comprised of Patients from 11 Centers.: 225 consecutive patients will be treated with local standard of care. The antiviral drug Tenofovir Disoproxil Fumarate (TDF) will be used to treat highly viremic chronic hepatitis B mothers from the gestational week 24-28 of pregnancy to delivery of infant at eleven centers across the People's Republic of China (PRC). Infants will receive hepatitis B vaccine plus HBIg at birth (within 12 hours) and additional hepatitis B vaccine at the age of week 4 and week 24.
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300mg for arm (B)

INTERVENTIONS:
Drug: Tenofovir Alafenamide 25 MG for arm (A) — Tenofovir Alafenamide (TAF) will be provided, 25 mg Per Oral daily.
  Other Names: HBIg 200 IU im for infants; HBV vaccine 10 ug im for infants
  Groups: Arm (A) TAF Group Comprised of Patients from 11 Centers.
Drug: Tenofovir Disoproxil Fumarate 300mg for arm (B) — Tenofovir Disoproxil Fumarate (TDF) will be provided, 300 mg Per Oral daily.
  Other Names: HBIg 200 IU im for infants; HBV vaccine 10 ug im for infants
  Groups: Arm (B) TDF Group Comprised of Patients from 11 Centers.

SUMMARY:
Immunoprophylaxis failure of hepatitis B (HBV) remains a concern and has been reported in approximately 10-30% of infants born to highly viremic mothers with HBeAg-positive. Maternal HBV DNA >6log10 copies/mL (or 200,000 IU/mL) is the major independent risk for mother-to-child transmission (MTCT). Two recent random controlled trial (RCT) studies have shown that the use of Tenofovir Disoproxil Fumarate (TDF) in highly viremic HBsAg positive mothers may safely reduce the rate of MTCT when compared between groups of TDF treated and untreated patients. Tenofovir Alafenamide (TAF) is the successor to TDF, and both drugs have a similar mechanism of action to reduce HBV DNA levels and normalize serum alanine aminotransferase (ALT) in chronic hepatitis B patients (CHB) with few adverse effects. TAF however, has a better safety profile with less adverse effects to bone mineral density and renal function. The present prospective, double-arm study is to evaluate the non-inferiority in the efficacy and safety of TAF therapy versus TDF therapy in highly viremic mothers and their infants for the prevention of MTCT in the real world setting.

DETAILED DESCRIPTION:
This is a prospective, double-arm, multi-center study conducted through 11 centers across China. Consecutive 450 mothers who are eligible for the study will be enrolled during gestational weeks 24-28 to receive TDF or TAF based on the patients' preference, and the treatment will be discontinued right after the delivery. All infants will receive HBV vaccination plus HBIg within 12 hours after birth and the additional HBV vaccination at the age of 4 weeks and 24 weeks. Primary outcome assessment will be performed at the infants' age of 28 will be collected to evaluate non-inferiority in the safety and efficacy of TAF therapy versus TDF therapy. These parameters will be extracted from test results of serum biochemistries, hematology, and virology, including but not limited to aspartate aminotransferase (AST), ALT, HBV DNA levels, and serological status of HBV (HBsAg, HBeAb, HBcAb, HBeAg, and HBsAg).

All aforementioned clinical parameters will be extracted from mothers at the following timepoints for assessment: the baseline, i.e. the start of TAF/TDF treatment, gestational weeks 28, 32, 36, on delivery, and at postpartum weeks 24-28. For the infant, information from two timepoints, at birth and at infant age of 28 weeks, will be collected. This information regarding the infant will include the physical parameters weight, height, head circumference, HBV DNA levels, HBV serological status, if they received hepatitis B immunoglobin (HBIg), if they received the complete series of HBV vaccine. All relevant information regarding the patient will be logged into a password-protected computer for primary and secondary analysis.

Group A: 225 participating mothers will receive TAF (oral 25 mg tablet daily) starting at gestational week 24-28 of pregnancy and continue until delivery. The mothers will be followed together with their infants until postpartum week 28.Infants will receive hepatitis B vaccine plus HBIg at birth (within 12 hours) and additional hepatitis B vaccine at the age of week 4 and week 24. Group B: 225 participating mothers will receive TDF (oral 300 mg tablet daily) starting at gestational week 24-28 of pregnancy and continue until delivery. Patients in group B will have similar follow-up schedules as those in the Group A. Infants will receive hepatitis B vaccine plus HBIg at birth (within 12 hours) and additional hepatitis B vaccine at the age of week 4 and week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant female, above 18 years of age and under 40 years of age.
2. Gestational age between 12-14 weeks (The screening on patients can be started at gestational week 12).
3. Documented compensated and stable chronic hepatitis B defined by all of the following:

   * HBsAg persistently positive > 6 months.
   * Clinical history, physical findings, and test results are compatible with compensated chronic hepatitis B.
4. Detectable maternal serum HBsAg and HBeAg at the screening visit.
5. Maternal serum HBV DNA levels exceeding 200,000 IU/mL by the COBAS Amplicor HBV PCR assay at screening visits.
6. Patient is willing and able to comply with the study drug regimen and all other study requirements. Patient is also willing to prevent another pregnancy in 28 weeks after delivery of the current baby.
7. Patient and her husband (both father and mother of the child) understand the risk and are willing to have the mother participating in the study. The mother must be willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

Patients will be excluded if they have any one of the following:

1. Creatinine clearance <100 mL/min (using the Cockcroft-Gault method based on serum creatinine and ideal body weight) or hypo-phosphoremia (below normal range).
2. History of renal events on adefovir or history of resistance to adefovir.
3. Hemoglobin <8 g/dL, or neutrophil count <1000/uL, or ALT >5 times ULN, or total bilirubin >2 mg/dL; or albumin <25gm/L, or abnormal creatinine level, or abnormal BUN levels.
4. History of abortion, or congenital malformation, or child infected with HBV in a prior pregnancy.
5. Biological father of the child (current pregnancy) has CHB.
6. Significant renal, cardiovascular, pulmonary, or neurological disease that may impact the subject's participation in the study as per the opinion of the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 225 consecutive chronically infected hepatitis B mothers who are willing to receive tenofovir alafenamide (TAF) treatment and another consecutive 225 who are willing to receive tenofovir disoproxil fumarate (TDF) treatment at eleven centers across China for high viremic load during pregnancy will be enrolled and followed prospectively for data collection. These patients underwent TAF/TDF treatment in their respective care centers and will be grouped together in Group A for TAF treatment and Group B for TDF treatment for primary and secondary analysis.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment on the Proportion of Infants who are Infected with Hepatitis B at the Age of 28 Weeks in the Two Groups | From the date of birth to the age of 24-28 weeks
  Compare MTCT rates between the two study groups and demonstrate non-inferiority in efficacy. MTCT rate is defined as the proportion of infants with serum HBV DNA >20 IU/mL and/or HBsAg positivity at 28 weeks of age.
Assessment on Congenital Defects and/or Malformation Rates in Each Infant Group for Comparison | from the date of birth to Infant's age of 24-28 weeks
  The rate of congenital defects and/or malformation rates in infants. Congenital defects and/or malformation rates are defined as the proportion of infants with the aforementioned abnormalities discovered during the study period. The rate of infant congenital defect/malformation as determined in group A will be compared with that of group B.

SECONDARY OUTCOMES:
Assessment on the change in Maternal HBV DNA Levels at Delivery | from gestational week 24-28 week to delivery
  Assess the change in maternal HBV DNA levels (IU/mL) at delivery when compared to the baseline before initiating TAF/TDF.
Maternal Serological Outcomes During the Study: Percentage of Mothers who Loss/Seroconversion of HBsAg or/and HBeAg During the Study | from gestational week 24-28 week to postpartum week 28
  Assess the percentage of mothers who loss/seroconversion of HBsAg or/and HBeAg during the study. Loss is defined by a test showing a negative HBsAg/HBeAg result at the end of the trial, given a positive respective test result at baseline. A seroconversion is defined as a test showing a negative HBsAg and a positive HBsAb result, or a negative HBeAg and a positive HBeAb result at the end of the trial, given a positive HBsAg/HBeAg test result at baseline. The proportion of mothers who experience loss/seroconversion as determined in group A will be compared with that of group B.
Incidence of Treatment-Emergent Adverse Events in Mothers as Stratified by the CTCAE v 5.0 | Gestational week 24-28 until Postpartum Week 28
  Assess the percentage of Mothers who have adverse events during the study, graded by the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. The proportion of mothers who experience adverse events as determined in group A will be compared with that of group B.
Incidence of Treatment-Emergent Adverse Events in Infants as Stratified by the CTCAE v 5.0 | Delivery until Infant age Week 28
  Assess the percentage of infants who have adverse events during the study, graded by the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. The proportion of infants who experience adverse events as determined in group A will be compared with that of group B.
Percentage of Mothers with Alanine transferase (ALT) Levels Within the Normal Limit | Gestational week 24-28 until Postpartum week 28
  To calculate the percentage of mothers at postpartum 28 weeks whose ALT (U/L) levels stay within the normal limit in response to therapy. The proportion of mothers whose ALT levels who stay within the normal limit as determined in group A will be compared with that of group B.
Percentage of Mothers with Aspartamine transferase (AST) Levels Within the Normal Limit | Gestational week 24-28 until Postpartum week 28
  To calculate the percentage of mothers at postpartum 28 weeks whose AST (U/L) levels stay within the normal limit in response to therapy. The proportion of mothers whose AST levels who stay within the normal limit as determined in group A will be compared with that of group B.
Group A: Proportion of Infants Born to Mothers Who Received TAF, Whose Physical Growth Characteristics Stay Within the Published National Normal Range. | Delivery to Infant age 28 weeks
  Physical growth characteristics of the infants, born to mothers who received TAF, at the time points on birth and infant age of 24-28 weeks will be compared with the normal range of the national database published in recent years and analyzed. The proportion of infants whose growth characteristics are outside the published national range at the end of the study as determined in group A will be compared with that of group B.
Group B: Proportion of Infants Born to Mothers Who Received TDF, Whose Physical Growth Characteristics Stay Within the Published National Normal Range. | Delivery to Infant age 28 weeks
  Physical growth characteristics of the infants, born to mothers who received TDF, at the time points on birth and infant age of 24-28 weeks will be compared with the normal range of the national database published in recent years and analyzed.The proportion of infants whose growth characteristics are outside the published national range at the end of the study as determined in group A will be compared with that of group B.
Tolerability of TDF vs TAF Therapy: Percentage of Mothers who Discontinue Therapy Due to the Adverse Event(s) During the Study. | Gestational week 24-28 until Delivery
  Assess the percentage of mothers who discontinue therapy due to the adverse event(s) during the study. The proportion of mothers who discontinue therapy as determined in group A will be compared with that of group B.

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Pan, MD, Principal Investigator — Beijing Ditan Hospital, Capital Medical University; NYU Langone Health, NY, USA
Locations (11):
- China (11):
  - Pingdingshan Hospital of Chongqing Public Health Medical Treatment Center, Shapingba, Chongqing Municipality
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Seventh Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The Third Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilonjiang
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Ganzhou Fifth People's Hospital, Ganzhou, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Public Health Clinical Center, Fudan University, Zhujing, Shanghai Municipality
  - Yuyao People's Hospital of Zhejiang Province, Yuyao, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xu WM, Cui YT, Wang L, Yang H, Liang ZQ, Li XM, Zhang SL, Qiao FY, Campbell F, Chang CN, Gardner S, Atkins M. Lamivudine in late pregnancy to prevent perinatal transmission of hepatitis B virus infection: a multicentre, randomized, double-blind, placebo-controlled study. J Viral Hepat. 2009 Feb;16(2):94-103. doi: 10.1111/j.1365-2893.2008.01056.x. Epub 2008 Oct 8. PMID 19175878
- [Background] Zou H, Chen Y, Duan Z, Zhang H. Protective effect of hepatitis B vaccine combined with two-dose hepatitis B immunoglobulin on infants born to HBsAg-positive mothers. PLoS One. 2011;6(10):e26748. doi: 10.1371/journal.pone.0026748. Epub 2011 Oct 28. PMID 22053208
- [Background] Pan CQ, Duan Z, Dai E, Zhang S, Han G, Wang Y, Zhang H, Zou H, Zhu B, Zhao W, Jiang H; China Study Group for the Mother-to-Child Transmission of Hepatitis B. Tenofovir to Prevent Hepatitis B Transmission in Mothers with High Viral Load. N Engl J Med. 2016 Jun 16;374(24):2324-34. doi: 10.1056/NEJMoa1508660. PMID 27305192
- [Background] Jourdain G, Ngo-Giang-Huong N, Harrison L, Decker L, Khamduang W, Tierney C, Salvadori N, Cressey TR, Sirirungsi W, Achalapong J, Yuthavisuthi P, Kanjanavikai P, Na Ayudhaya OP, Siriwachirachai T, Prommas S, Sabsanong P, Limtrakul A, Varadisai S, Putiyanun C, Suriyachai P, Liampongsabuddhi P, Sangsawang S, Matanasarawut W, Buranabanjasatean S, Puernngooluerm P, Bowonwatanuwong C, Puthanakit T, Klinbuayaem V, Thongsawat S, Thanprasertsuk S, Siberry GK, Watts DH, Chakhtoura N, Murphy TV, Nelson NP, Chung RT, Pol S, Chotivanich N. Tenofovir versus Placebo to Prevent Perinatal Transmission of Hepatitis B. N Engl J Med. 2018 Mar 8;378(10):911-923. doi: 10.1056/NEJMoa1708131. PMID 29514030
- [Background] Wiseman E, Fraser MA, Holden S, Glass A, Kidson BL, Heron LG, Maley MW, Ayres A, Locarnini SA, Levy MT. Perinatal transmission of hepatitis B virus: an Australian experience. Med J Aust. 2009 May 4;190(9):489-92. doi: 10.5694/j.1326-5377.2009.tb02524.x. PMID 19413519